CLINICAL TRIAL: NCT01504958
Title: Effects of a Combined TMS and Cognitive Training in Alzheimer Patients: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Effects of a Combined Transcranial Magnetic Stimulation (TMS) and Cognitive Training in Alzheimer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Neuronix Ltd (Industry)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010P000325
Record Dates: First submitted 2011-09-29; First posted 2012-01-06 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; Cognitive Training; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Alzheimer Disease | interventions — Transcranial Magnetic Stimulation; Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active rTMS with real cognitive training (Active Comparator): High frequency rTMS stimulation to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area) paired with concurrent active cognitive training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: NICE Cognitive Training
- Sham rTMS with real cognitive training (Sham Comparator): High frequency sham rTMS to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area) paired with concurrent active cognitive training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: NICE Cognitive Training
- Sham rTMS with sham cognitive training (Sham Comparator): High frequency sham rTMS to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area) paired with concurrent sham cognitive training.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS); Behavioral: NICE Cognitive Training

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — Each subject will receive up to 1800 pulses of up to 20Hz per day to all simulated brain regions together. Treated brain areas will be alternated each day (only 3 a day).
  Sham participants will receive the same study procedures as patients receiving active rTMS.
  Other Names: Transcranial Magnetic Stimulation; Noninvasive Brain Stimulation
Behavioral: NICE Cognitive Training — 12 levels of difficulty in tasks designed to relate to the region of the brain being stimulated (left and right parietal cortex, left and right DLPFC, left superior temporal gyrus, left inferior frontal gyrus).
  A particular cognitive exercise will start 200msec after the termination of each TMS train.
  Sham participants receive sham cognitive training that follows the same procedures as the active group.
  Other Names: Cognitive Training; Mental exercises

SUMMARY:
This study looks at the potential benefits of combining cognitive training (mental exercises) together with transcranial magnetic stimulation (also known as TMS) to see if this can make a difference in the condition of people with Alzheimer's disease by improving their disease and the cognitive decline that goes along with it.

DETAILED DESCRIPTION:
This study takes place in Boston, Massachusetts and Beth Israel Deaconess Medical Center. The treatment portion of the study requires patients to visit the BIDMC daily, Monday through Friday, for 6 weeks. All participants will receive real cognitive training, but half of our participants will receive active TMS treatment and half will receive a placebo TMS treatment. However, those receiving the placebo treatment will be offered the real treatment upon the completion of the study. This study goes up to approximately 4.5 months.

TMS is a noninvasive way of stimulating the brain, which is not painful and does not involve any needles or any form of surgery. It acts by delivering a magnetic stimulation to a particular region of your brain and that, coupled with the cognitive training, is what is being looked at in this study. The investigators are examining if this combination of TMS and cognitive training will improve your memory function and other mental functions such as language, orientation, and thinking or judgment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 55-90
* Diagnosed with mild to moderate AD according to DSM-IV criteria
* Diagnosis of dementia of the Alzheimer's type according to the criteria established by the NINCDS-ADRDA
* Normal or corrected normal ability to see and hear
* Primary language is English

Exclusion Criteria:

* IQ below 85
* Any major structural abnormalities on MRI (eg. Infarction, intracerebral malformation)
* Any symptoms of disease or abnormalities sufficient to cause memory impairment other than AD (eg. Normal pressure hydrocephalus, progressive supranuclear palsy)
* Any functional psychiatric disorder (eg. Schizophrenia)
* Chronic uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (eg. Cardiac malformation)
* History of seizures, diagnosis of epilepsy
* Metal implants excluding dental fillings or any of the following medical devices: pacemaker, implanted medication pump, vagal nerve stimulator, deep brain stimulator, TENS unit (unless removed completely for this study), cerebral spinal fluid shunt
* Recent withdrawal from the following drugs: alcohol, barbiturates, benzodiazepines, meprobamate, chloral hydrate

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, M.D., Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Bentwich J, Dobronevsky E, Aichenbaum S, Shorer R, Peretz R, Khaigrekht M, Marton RG, Rabey JM. Beneficial effect of repetitive transcranial magnetic stimulation combined with cognitive training for the treatment of Alzheimer's disease: a proof of concept study. J Neural Transm (Vienna). 2011 Mar;118(3):463-71. doi: 10.1007/s00702-010-0578-1. Epub 2011 Jan 19. PMID 21246222
- [Derived] Brem AK, Di Iorio R, Fried PJ, Oliveira-Maia AJ, Marra C, Profice P, Quaranta D, Schilberg L, Atkinson NJ, Seligson EE, Rossini PM, Pascual-Leone A. Corticomotor Plasticity Predicts Clinical Efficacy of Combined Neuromodulation and Cognitive Training in Alzheimer's Disease. Front Aging Neurosci. 2020 Jul 8;12:200. doi: 10.3389/fnagi.2020.00200. eCollection 2020. PMID 32733232
- See also: Related Information to the Alzheimer's Trial; sponsors website. — http://www.neuronixmedical.com/neuroAD/
- See also: Related Information regarding the TMS lab at Beth Israel Deaconess Medical Center — http://tmslab.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Active rTMS With Real Cognitive Training: High frequency rTMS stimulation to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area).
  Repetitive Transcranial Magnetic Stimulation (rTMS): Each subject will receive up to 1800 pulses of up to 20Hz per day to all simulated brain regions together. Treated brain areas will be alternated each day (only 3 a day).
  Sham participants will receive the same study procedures as patients receiving active rTMS.
  NICE Cognitive Training: 12 levels of difficulty in tasks designed to relate to the region of the brain being stimulated (left and right parietal cortex, left and right DLPFC, left superior temporal gyrus, left inferior frontal gyrus).
  A particular cognitive exercise will start 200msec after the termination of each TMS train.
  Sham participants receive real cognitive training that follows the same procedures as the active group.
- Sham rTMS With Real Cognitive Training: High frequency sham rTMS to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area).
  Repetitive Transcranial Magnetic Stimulation (rTMS): Each subject will receive up to 1800 pulses of up to 20Hz per day to all simulated brain regions together. Treated brain areas will be alternated each day (only 3 a day).
  Sham participants will receive the same study procedures as patients receiving active rTMS.
  NICE Cognitive Training: 12 levels of difficulty in tasks designed to relate to the region of the brain being stimulated (left and right parietal cortex, left and right DLPFC, left superior temporal gyrus, left inferior frontal gyrus).
  A particular cognitive exercise will start 200msec after the termination of each TMS train.
  Sham participants receive real cognitive training that follows the same procedures as the active group.
- Sham rTMS With Sham Cognitive Training: High frequency sham rTMS stimulation to the left and right parietal cortex (somatosensory association cortex), left and right DLPFC (dorsolateral prefrontal cortex), and left superior temporal gyrus (Broca's area).
  Repetitive Transcranial Magnetic Stimulation (rTMS): Each subject will receive up to 1800 pulses of up to 20Hz per day to all simulated brain regions together. Treated brain areas will be alternated each day (only 3 a day).
  Sham participants will receive the same study procedures as patients receiving active rTMS.
  Sham Cognitive Training: subjects will undergo pseudo cognitive training with the sham rTMS following the same procedures as the active group
Period: Overall Study
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training
Started | 10 (Baseline clinical, cognitive, and behavioral assessments: TMS-EMG measures, MRI scan, randomization.) | 6 (Baseline clinical, cognitive, and behavioral assessments: TMS-EMG measures, MRI scan, randomization.) | 6 (Baseline clinical, cognitive, and behavioral assessments: TMS-EMG measures, MRI scan, randomization.)
Completed | 10 (1 Month Post-Treatment Follow Up) | 6 (1 Month Post-Treatment Follow Up) | 6 (1 Month Post-Treatment Follow Up)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number analyzed: 21 (1 enrolled was excluded from analysis) Real/Real: 10 Real/Sham: 5 Sham/Sham: 6
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training | Total
Number analyzed (Participants) | 10 | 5 | 6 | 21
Age, Continuous [Mean (Full Range); unit: years] | 69.1 [52 to 76] | 68.6 [54 to 86] | 70 [54 to 86] | 69.24 [52 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 2 | 12
  Male | 3 | 2 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)
Description: Assessment to measure the severity of all of the most important symptoms of Alzheimer's disease: loss of memory, language, praxis, and attention. The total scoring range is 0-70, with 0 representing the least impairment and 70 the most severe impairment. The results posted below represent a change in score from baseline. A positive change represents an improvement on the ADAS-Cog (change = 1 month score - baseline score).
Time Frame: Pre treatment; 1 month post treatment
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training
Number analyzed (Participants) | 10 | 5 | 6
percentage change | 1.79 (3.60) | -0.20 (5.45) | -0.66 (2.91)

2. Secondary Outcome: Clinical Global Impression of Change (CGIC)
Description: The CGI is a three-item scale used to assess treatment response in psychiatric patients. The CGI-C subset measures the global improvement or change from baseline. Scores range from 0 to 7, with 0 indicating marked improvement and 7 indicating marked worsening. The scores below represent the percent change of the scores from baseline.
Time Frame: Pre-treatment, 1 month post treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training
Number analyzed (Participants) | 10 | 5 | 6
percent change | 3.25 (0.72) | 4.40 (0.89) | 4.08 (1.02)

3. Secondary Outcome: Alzheimer's Disease Cooperative Study - Activities of Daily Living Inventory (ADCS-ADL)
Description: 23 item scale to assess activities of daily living. Scores range from 0 to 78 with a higher score indicating less functional impairment. The scores reported below are the means of the actual scores from the assessments representing the percent change from baseline.
Time Frame: Pre-treatment, 1 month Post-treatment
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training
Number analyzed (Participants) | 10 | 5 | 6
percent change
  Pre-Treatment | 72.67 (5.07) | 73.60 (3.36) | 65.75 (6.80)
  Post-Treatment | 69.78 (7.80) | 71.20 (5.93) | 61.75 (9.50)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to 1 month post-treatment
Description: All adverse events were self-reported according to a Side Effects Questionnaire administered at each visit.
Arm/Group | Active rTMS With Real Cognitive Training | Sham rTMS With Real Cognitive Training | Sham rTMS With Sham Cognitive Training
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 5/10 | 5/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active rTMS With Real Cognitive Training (N=10) | Sham rTMS With Real Cognitive Training (N=6) | Sham rTMS With Sham Cognitive Training (N=6)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — A subject sustained a 5cm contusion and subtle rib fracture resulting from a fall at home. Subject was brought to the hospital for evaluation. Subject was in the follow up phase. This was assessed as unlikely related to to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active rTMS With Real Cognitive Training (N=10) | Sham rTMS With Real Cognitive Training (N=6) | Sham rTMS With Sham Cognitive Training (N=6)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — Subject experienced twitching in bicep and wrist flexor of the right arm at the beginning of a TMS session that lasted for 5 seconds and resolved. Subject also reported nausea and session was discontinued.
Headache (Nervous system disorders) | 5 | 5 | 0 — Reported headaches ranged from mild to moderate post-intervention as compared to pre-intervention. Most were assessed as possibly/probably related to the study.
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 — Reported mild neck pain/stiffness post-intervention.
Scalp Pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 — Reported mild scalp pain post-intervention
Hearing Impairment (Ear and labyrinth disorders) | 1 | 1 | 0 — Reported mild hearing impairment post-intervention as compared to pre-intervention. Earplugs were worn throughout every session. No long term hearing impairment reported.
Impaired Cognition (Nervous system disorders) | 0 | 1 | 0 — Reported mild impaired cognition post-intervention compared to pre-intervention. Most reported as tiredness. No long term impairment reported.
Trouble Concentrating (Nervous system disorders) | 0 | 4 | 0 — Reported mild trouble concentrating post-intervention as compared to pre-intervention. Most reported as tiredness. No long term trouble reported.
Tiredness (Nervous system disorders) | 3 | 1 | 0 — Reported mild tiredness post-intervention as compared to pre-intervention.
Soreness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Participant reported mild soreness at the inferior frontal gyrus (stimulation site) post-stimulation.
Blurry Vision (Eye disorders) | 1 | 0 | 0 — Blurry vision reported after looking at computer screen for extended period of time
Anxiousness (Psychiatric disorders) | 1 | 1 | 0 — Reported increase in anxiety post-intervention
Dizziness (Nervous system disorders) | 1 | 1 | 0 — Reported mild dizziness post-intervention as compared to pre-intervention.
Depression (Psychiatric disorders) | 0 | 1 | 0 — Participant reported feeling mildly subdued/dazed/depressed following intervention. No long term effects.
Achiness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Reported mild achiness post-intervention.
Muscle Heaviness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Reported mild eye heaviness post-intervention. No long term effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No